CLINICAL TRIAL: NCT04950478
Title: THE EFFECT OF VIRTUAL REALITY ON PAIN EXPERIENCED BY SCHOOL-AGE CHILDREN DURING VENIPUNCTURE: RANDOMIZED CONTROLLED STUDY
Brief Title: Effect of Virtual Reality on Child Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eda Orhan, PhD RN, Educator Nurse, Koc University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Virtual Reality use on Pain
Record Dates: First submitted 2021-06-29; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Pain
Keywords: child; nursing; pain management; venipuncture; Virtual reality
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The children wore the virtual reality headset and game was started one minute before the venipuncture. The children took off the virtual reality headset after the venipuncture ended.
  Interventions: Other: Virtual Reality
- Control Group (No Intervention): No intervention was performed to reduce pain in the control group

INTERVENTIONS:
Other: Virtual Reality — 5 minutes before the procedure, they were recorded on 'Child and Parent Information Form', State-Trait Anxiety Inventory for Children and FPS-R. Their heart rate and oxygen saturation values were read and recorded. Children wore the virtual reality headset and game was started one minute before the venipuncture. As soon as the injector inserted, the researcher turned on a stopwatch and read and recorded heart rate and oxygen saturation values. When the injector was removed, the researcher stopped the stopwatch and recorded the duration of the procedure.When the injector was removed, the stopwatch was stopped and heart rate and oxygen saturation were recorded. The children took off the virtual reality headset and were asked to evaluate their pain level through FPS-R and their responses were recorded.
  Arms: Virtual Reality

SUMMARY:
This study is a randomized controlled experimental study conducted to determine effect of using virtual reality headset during venipuncture on pain level, heart rate and oxygen saturation values among 7-12 year-old children. The data were collected from 102 children coming to vaccination room of an university hospital's pediatric outpatient clinic. Before the venipuncture, state anxiety scores of children in both groups were evaluated. The children in experimental group wore virtual reality headset during the venipuncture. The children in control group were subjected to standard venipuncture procedure. Before, during and after the venipuncture, pulse and oxygen saturation values were measured.

DETAILED DESCRIPTION:
The research was designed as a randomized controlled experimental study. The population of the study consisted of all 7-12 year-old children who came to a vaccination room of an university hospital's pediatric outpatient clinic .It is stated in the literature that the sample size should be determined as minimum 41 in both experimental and control groups in the experimental studies.

In the study, randomization Urn method was carried out. Urn method consists of two parameters (α and β). These parameters are matched with two different colored balls (red and white). One of the balls was randomly selected and if this ball was white, the individual was assigned to α group; if it was red, then participant was assigned to β group. This process was repeated for each assignment. In the study, white ball was determined as control group; whereas, red ball was determined as experimental group. In the case of a child meeting the sampling criteria, these balls that the researcher had previously prepared were placed in a black bag and any nurse working in the pediatrics outpatient clinic at that time was asked to draw a ball from the bag. The children were assigned to experimental or control group based on color of the selected ball so that they were randomly distributed to two groups. A total of 106 children including 54 children in the experimental group and 52 children in the control group were included in the sample group by taking possible case losses into account. Since 2 children in the experimental group did not want to wear the virtual reality headset during the procedure, they were excluded from the sample. 2 children in the control group were excluded from the sample because venipuncture procedure did not take place at once. Thus, the sample group consisted of 102 children in total including 52 children in the experimental group and 50 children in the control group. The study followed the CONSORT guideline for reporting randomized controlled trials. The data collection questionnaries included a Child and Parent Information Form, State-Trait Anxiety Inventory for Children, and Faces Pain Scale-Revised (FPS-R).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12 who agreed to participate in the study by giving written and verbal consent,
* Parents who agreed to participate in the study verbally and in written by signing informed consent form,
* Body temperature within normal values for children (36.5- 37.2 oC),
* Children who were healthy and for whom the doctor requested a blood test for general control.
* Children who were healthy in sensory and neurologic aspects.

Exclusion Criteria:

* Having any chronic disease or any disease causing pain in children,
* Having hearing, mental or neurological disability in children,
* Having history of syncope during previous venipuncture procedures for the children,
* Having visual impairment in children,
* Unsuccessful venipuncture procedure in the first attempt.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Between 5-10 minutes
  The children were informed about the Faces Pain Scale-Revised (FPS-R) and they were asked to mark the children's pain levels on the scale before and after the venipuncture procedure. In addition, the pain levels of the children before and after the procedure were determined by the researcher who is a specialist in pediatric nursing by using the same scales.

SECONDARY OUTCOMES:
Heart Rate | Between 5-10 minutes
  Heart rate values were read and recorded form the pulse oximeter before venipuncture, as soon as the injector inserted and after the injector removed.
Oxygen Saturation | Between 5-10 minutes
  Oxygen saturation values were read and recorded form the pulse oximeter before venipuncture, as soon as the injector inserted and after the injector removed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa Florence Nightingale Faculty of Nursing, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Orhan E, Gozen D. The Effect of Virtual Reality on Pain Experienced by School-Age Children During Venipuncture: A Randomized Controlled Study. Games Health J. 2023 Aug;12(4):330-339. doi: 10.1089/g4h.2022.0232. PMID 37466456